CLINICAL TRIAL: NCT02881697
Title: mTOR and Adipose Tissue Inflammation in Humans
Brief Title: mTOR and Adipose Tissue Inflammation
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: mTOR
Record Dates: First submitted 2016-08-18; First posted 2016-08-29 (Estimated); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Adipose tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Obese insulin-resistant subjects: Adipose tissue sampling in obese volunteers (BMI > 35kg/m2) aged 18- max. 60 years, males and females; insulin-resistant, scheduled for elective bariatric surgery
  Interventions: Other: Adipose tissue sampling
- Lean insulin-sensitive controls: Adipose tissue sampling in normal weight patients (BMI < 27kg/m2) aged 18- max. 60 years, males and females; insulin-sensitive, scheduled for elective surgery
  Interventions: Other: Adipose tissue sampling
- Obese diabetic subjects: Adipose tissue sampling in obese volunteers (BMI > 35kg/m2) aged 18- max. 60 years, males and females; diabetic, scheduled for elective bariatric surgery
  Interventions: Other: Adipose tissue sampling

INTERVENTIONS:
Other: Adipose tissue sampling

SUMMARY:
The target of rapamycin complex 2 (TORC2) is an evolutionarily conserved serine/threonine protein kinase that controls growth and metabolism. In mammals (including humans), mammalian TOR complex 2(mTORC2) contains mammalian TOR (mTOR), RICTOR, mSIN1 protein, and mLST8 gene. In an animal model, the adipose-specific rictor knockout (AdRiKO) mouse, systemic insulin resistance, hepatic steatosis, and cardiovascular dysfunction develop upon high fat diet (HFD)-induced obesity or aging. To find a molecular link between adipose mTORC2 and systemic insulin resistance, investigators have already performed transcriptomics and proteomics analysis on visceral white adipose tissue in a mouse model. The aim of the study is to confirm a molecular link between adipose mTORC2 and systemic insulin resistance in humans.

ELIGIBILITY:
Inclusion Criteria:

* Obese volunteers (BMI > 35kg/m2) aged 18 to a maximum of 60 years, males and females; insulin-resistant, scheduled for elective bariatric surgery.
* Normal weight patients (BMI < 27kg/m2) aged 18- max. 60 years, males and females; insulin-sensitive, scheduled for elective surgery.

Exclusion Criteria:

* Known diabetes mellitus
* Chronic inflammatory disease (inflammatory bowel disease, rheumatoid disease, cancer)
* Acute inflammatory disease
* Known renal disease: kidney failure
* Pregnancy:
* history of gastrointestinal surgery with major changes to the gastrointestinal tract (removal of stomach, any GI-bypass)
* Substance abuse, alcohol abuse
* Inability to follow procedures due to psychological disorders, dementia
* insufficient knowledge of project language (German)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Obese patients (BMI >35 kg/m2) with insulin resistance and lean controls (BMI < 27kg/m2) scheduled for elective surgery for non-inflammatory conditions such as gallstone disease, diverticular disease or - in the case of obese subjects - bariatric surgery
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2016-09-27 (Actual); Primary Completion 2019-04-23 (Actual); Study Completion 2019-07-27 (Actual)

PRIMARY OUTCOMES:
mTORC2 activity in adipose tissue measured by immunoblot | single time point at surgery
  measurement of mTORC2 activity in adipose tissue once at surgery

SECONDARY OUTCOMES:
Mcp1 messenger ribonucleic acid (mRNA) level in adipose tissue measured by quantitative polymerase chain reaction (PCR) | single time point at surgery
  measurement of Mcp1 messenger ribonucleic acid (mRNA) level in adipose tissue once at surgery

OTHER OUTCOMES:
Insulin resistance measured with fasting plasma insulin and fasting glucose | single time point at surgery
  measurement of fasting plasma insulin and fasting Glucose once at surgery

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Beglinger, MD, Study Chair — St. Claraspital klinische Forschungsabteilung

IPD SHARING:
Plan to Share IPD: Undecided